CLINICAL TRIAL: NCT01987180
Title: NICU-2-HOME: Using HIT to Support Parents of NICU Graduates Transitioning Home
Brief Title: Using Smartphones in the Neonatal Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Craig Garfield, Associate Professor, Northwestern University
Other Study IDs: NICU2Home Feasability
Record Dates: First submitted 2013-10-31; First posted 2013-11-19 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Self-efficacy
Keywords: self-efficacy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Usual standard care: Parents will be provided with the usual standard of care in the NICU. Discharge information will be provided to parents as is typically done in the NICU for VLBW infants getting ready to go home. Typical handouts are given to parents that describe their child's care and needs specifically as well as general guidelines. The project coordinator for the research study will verify that parents received information prior to discharge from the NICU staff. Parents will determine how you use this information.
- NICU-2-Home mobile app user: Parents will receive smartphone and unique NICU-2-Home app for their use. A pair of parents will be given two smartphones and will be asked to use the devices in their preferred way. Within the given app there is a baby tracking tool (baby-connect.com) that enables parents to keep track of the baby's feeding, diapers, sleep, health, medicines, vaccines, photos, etc. The objective in doing this is not to monitor the growth and development of the child; rather, it is to observe what tools within the app parents use and how frequently they use them.

SUMMARY:
The goal of this research is to develop and pilot the NICU-2-Home service, a health information technology (IT) concept centered on a smart phone app. NICU-2-Home will provide support to parents of very low birth weight (VLBW) infants as they transition from the NICU to their homes and eventually establish a medical home with the infant's pediatrician. Once the app is developed, we will conduct a feasibility study with randomization to pilot test the ability of NICU-2-Home app to (a) improve parent's self-efficacy and confidence in caring for their VLBW infant, (b) decrease parental stress, and (c) enhance involvement with their VLBW infants compared to controls.

DETAILED DESCRIPTION:
After 2-3 months in the Neonatal Intensive Care Unit (NICU), mothers and fathers of Very Low Birth Weight (VLBW) infants face discharge home with trepidation. Having a VLBW infant that has survived to discharge, these parents now must perform a myriad of health care tasks once at home, yet parents often feel ill-prepared, uninformed, and unskilled to provide this care. The goal of this exploratory research is to develop and pilot the NICU-2-Home service, a health information technology (IT) concept centered on the smart phone that will be created with researchers at Motorola. NICU-2-Home will provide support to parents of VLBW infants as they transition from the NICU to their homes and eventually establish a medical home with the infant's pediatrician. Phase 1 of this research uses qualitative methods and an iterative process to design the NICU-2-Home content service that will support parents as they transition to home from the NICU through interviews with the major stakeholders: parents, neonatal physicians, neonatal staff, and community pediatricians. Phase 2 evaluates NICU-2-Home as parents are transitioning to home and includes a feasibility study with randomization to pilot test the ability of NICU-2-Home to (a) improve parent's self-efficacy and confidence in caring for their VLBW infant, (b) decrease parental stress, and (c) enhance involvement with their VLBW infants compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Older than 18 years old
* Have at least one VLBW infant who survived to discharge and transitioned to home

Exclusion Criteria:

- N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of Very Low Birth Weight infants preparing for transition to home
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
saliva collection | 2 weeks before discharge and 2 weeks after discharge
  Parents will be asked to provide saliva samples at four different days (the day prior to discharge, the day after discharge, five days after discharge, and 2 weeks after discharge) at the following three times each day: when they wake up, 30 minutes later, and at bedtime.

SECONDARY OUTCOMES:
Questionnaires to measure change from baseline in parents' distress and depression | 2 weeks before discharge (baseline) and 2 weeks after discharge
  Parents will be asked to complete a particular set of surveys depending on which study day they are on. The study days include: 2 weeks prior to discharge (baseline), the day prior to discharge, the day after discharge, five days after discharge, and 2 weeks after discharge. Parents will complete the surveys independently without consulting their partner.
  The survey includes parenting sense of competence scale (PSOC), revised dyadic adjustment scale (RDAS), edinburgh postnatal depression scale (EPDS),perceived stress scale (PSS)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Garfield, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States